CLINICAL TRIAL: NCT05289531
Title: Validation of the Turkish Translation of the Low Anterior Resection Syndrome (LARS) Score
Brief Title: (LARS) Score Validation of Turkish Language
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Collaborators: Aarhus University Hospital (Other); Dokuz Eylul University (Other); Lokman Hekim University (Other Government)
Responsible Party: Principal Investigator, I Ethem Gecim, Professor of Surgery, Ankara University
Other Study IDs: 3
Record Dates: First submitted 2022-02-17; First posted 2022-03-21 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: LARS - Low Anterior Resection Syndrome
Keywords: Turkish LARS
MeSH Terms: conditions — Low Anterior Resection Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Rectal resection patients: Four Turkish centers participated in data collection in 2016. The inclusion criteria were rectal adenocarcinoma within 15 cm from the anal verge and LAR with either PME or TME. All patients had bowel continuity restored for at least 18 months when invited for the study. Exclusion criteria included failed R0 surgery, recurrence or dissemination, having intestinal stoma, previous cancer (except minor skin cancers) dementia and inability to speak Turkish (i.e., the need for a translator during treatment). A research assistant at each center identified the consecutive series of eligible patients for each participating consultant surgeon
  Interventions: Procedure: Rectal Resection Patients
- 52 patients re-questioned to answer the same questionaire as control group: The test-retest reliability of the LARS score was evaluated by asking 52 randomly selected subgroup of eligible patients to repeat the assessment of the LARS score 2 to 4 weeks after their initial response. Agreement between tests for the LARS score category and for each of the five LARS score items is presented as proportions with 95% confidence intervals. We considered it a perfect agreement if the patient ticked the exact same response category at both tests, a moderate agreement if responses differed by one category, while 'no agreement' was applied to patients whose responses differed by two or more categories.
  The intraclass correlation coefficient was used to evaluate the agreement between the initial test and the retest. The limit of agreements was calculated by using the Bland-Altman method. An ICC between 0.61 and 0.80 is considered strong agreement. A "p value" less than 0.05 was considered significant.
  Interventions: Procedure: Rectal Resection Patients

INTERVENTIONS:
Procedure: Rectal Resection Patients — Patients who have had low anterior resection of rectum was categorized for their quality of life related to surgery

SUMMARY:
Long-term bowel dysfunction after resection for rectal cancer, known as low anterior resection syndrome (LARS), is observed in many patients. The LARS score was developed to measure this syndrome and its impact on quality of life in Danish patients. Recently, English and many other language versions have been validated. The aim of this study was to validate the Turkish translation of the LARS score in Turkish patients who have undergone treatment for rectal cancer.

DETAILED DESCRIPTION:
A total of 326 patients were reviewed and contacted for the study, and 222 (68%) were eligible for the analyses. The association between the LARS score and quality of life and the test-retest reliability were studied. The intraclass correlation coefficient (ICC) was calculated to understand the degree of reliability.

ELIGIBILITY:
Inclusion Criteria:The inclusion criteria were

* rectal adenocarcinoma within 15 cm from the anal verge
* LAR with either PME or TME.
* Bowel continuity restored for at least 18 months when invited for the study.

Exclusion Criteria:Exclusion criteria included

* failed R0 surgery,
* recurrence or dissemination,
* having intestinal stoma,
* previous cancer (except minor skin cancers)
* dementia and inability to speak Turkish (i.e., the need for a translator during treatment).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients had their surgeries performed by expert colorectal surgeons with at least 15 years of experience and performing more than 20 rectal cancer surgeries in a year to minimize surgeon-related hazards for poor functional outcome. The first rectal resection with a diverting ileostomy in the study group was performed in May 2000, which was closed in January 2001, and the last stoma closure was in September 2018. All patients had their bowel continuity restored for at least 6 months prior to completing the survey.
Sampling Method: Non-Probability Sample
Enrollment: 222 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Validity of LARS Score | From Feb 2016 to Feb 2020
  The translated questionaire was validated on Turkish speaking patients

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Celasin H, Akyol C, Gecim IE, Halil Elhan A, Juul T, Sokmen S, Sungurtekin U, Akyuz S. Validation of the Turkish translation of the low anterior resection syndrome (LARS) score. Tech Coloproctol. 2023 Jun;27(6):465-474. doi: 10.1007/s10151-023-02751-z. Epub 2023 Jan 18. PMID 36650405